CLINICAL TRIAL: NCT06004297
Title: Influence of Combined Double-Bundle ACL Reconstruction With Lateral Retinacular Release to Prevent Patellofemoral Malalignment in Isolated ACL Rupture: a Randomized Controlled Trial
Brief Title: Influence of Combined Double-Bundle ACL Reconstruction With Lateral Retinacular Release to Prevent Patellofemoral Malalignment in Isolated ACL Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ludwig Andre Pontoh, DR., dr., Sp.OT(K), Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP/2019/003
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Single bundle group
  Interventions: Procedure: ACL reconstruction
- Group 2 (Active Comparator): Double bundle only group
  Interventions: Procedure: ACL reconstruction
- Group 3 (Experimental): Double bundle with lateral release group
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — performed arthroscopically

SUMMARY:
Anterior knee pain which might be due to patellofemoral malalignment is an inevitable post operative complication after an ACL reconstruction (ACLR). We combined the double bundle ACLR technique with lateral release technique to prevent patellofemoral malalignment post ACLR.

ELIGIBILITY:
Inclusion Criteria:

* unilateral isolated total ACL rupture
* normal BMI

Exclusion Criteria:

* flexion contracture more than 200, presence of anterior knee pain before surgery, Q angle >140 in males and >170 in females, presence of a patellar tilting, rupture of other ligaments, and muscular dysfunction.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
TTTG value | 6 months
  tibial tuberosity to trochlea groove, radiographic outcome

SECONDARY OUTCOMES:
Kujala score | 6 months
  functional outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No